CLINICAL TRIAL: NCT00740870
Title: Implantation of the Medtronic Melody Transcatheter Pulmonary Valve in Patients With Dysfunctional Right Ventricular Outflow Tract (RVOT) Conduits: A Feasibility Study
Brief Title: Melody Transcatheter Pulmonary Valve Study: Post Approval Study of the Investigational Device Exemption Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G050186
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Defects; Dysfunctional Right Ventricular Outflow Tract Conduits
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melody TPV Implant (Experimental): Melody Transcatheter Pulmonary Valve implanted into a dysfunctional RVOT Conduit.
  Interventions: Device: Transcatheter Pulmonary Valve replacement

INTERVENTIONS:
Device: Transcatheter Pulmonary Valve replacement — Transcatheter valve implantation into a RVOT conduit in patients with complex congenital heart defects where the conduit has become dysfunctional and where the patient needs invasive intervention.
  Other Names: Melody Transcatheter Pulmonary Valve

SUMMARY:
The primary objective is to confirm the long-term functionality of implantation of the Medtronic Melody TPV at 5 years is no worse than the historical control established through literature review. The secondary objectives are to evaluate long-term functionality at 10 years and to assess safety, procedural success, and clinical utility of transcatheter implantation of the Melody TPV.

DETAILED DESCRIPTION:
The primary objective is to confirm the long-term functionality of implantation of the Medtronic Melody TPV at 5 years is no worse than the historical control established through literature review. The secondary objectives is to evaluate long-term functionality at 10 years and to assess safety, procedural success, and clinical utility of transcatheter implantation of the Melody TPV.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 5 years of age
* Weight greater than or equal to 30 kilograms
* Existence of a full (circumferential) RVOT conduit that was equal to or greater than 16 mm in diameter when originally implanted, or a stented bioprosthesis with a rigid circumferential sewing ring in the RVOT that has an internal diameter greater than or equal to 18 mm and less than or equal to 22 mm when originally implanted.
* Any of the following by transthoracic echocardiography:
* For patients in New York Heart Association (NYHA) Classification II, III, or IV: Moderate (3+) or severe (4+) pulmonary regurgitation AND/OR Mean RVOT gradient greater than or equal to 35 mmHg
* For patients in NYHA Classification I:Severe (4+) pulmonary regurgitation with RV dilatation or dysfunction AND/OR Mean RVOT gradient greater or equal to 40 mmHg

Exclusion Criteria:

* Active endocarditis
* Major or progressive non-cardiac disease (liver failure, renal failure, cancer)that has a life expectancy of less than one year
* Patient or guardian unwilling or unable to provide written informed consent or comply with follow-up requirements
* Obstruction of the central veins (including the superior and inferior vena cava, bilateral iliac veins) such that the delivery system cannot be advanced to the heart via transvenous approach from either femoral vein or internal jugular vein
* Positive urine or serum pregnancy test 24 hours prior to procedure in female patients of child bearing potential
* Known intravenous drug abuse

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of NY-Presbyterian, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Seattle Children's and Regional Hospital, Seattle, Washington

REFERENCES:
- [Derived] Jones TK, McElhinney DB, Vincent JA, Hellenbrand WE, Cheatham JP, Berman DP, Zahn EM, Khan DM, Rhodes JF Jr, Weng S, Bergersen LJ. Long-Term Outcomes After Melody Transcatheter Pulmonary Valve Replacement in the US Investigational Device Exemption Trial. Circ Cardiovasc Interv. 2022 Jan;15(1):e010852. doi: 10.1161/CIRCINTERVENTIONS.121.010852. Epub 2021 Dec 21. PMID 34930015
- [Derived] Armstrong AK, Berger F, Jones TK, Moore JW, Benson LN, Cheatham JP, Turner DR, Rhodes JF, Vincent JA, Zellers T, Lung TH, Eicken A, McElhinney DB. Association between patient age at implant and outcomes after transcatheter pulmonary valve replacement in the multicenter Melody valve trials. Catheter Cardiovasc Interv. 2019 Oct 1;94(4):607-617. doi: 10.1002/ccd.28454. Epub 2019 Aug 16. PMID 31419019
- [Derived] Priromprintr B, Silka MJ, Rhodes J, Batra AS. A prospective 5-year study of exercise performance following Melody valve implant. Am Heart J. 2019 Mar;209:47-53. doi: 10.1016/j.ahj.2018.12.014. Epub 2018 Dec 29. PMID 30682562
- [Derived] Priromprintr B, Silka MJ, Rhodes J, Batra AS. A prospective 5-year study of the frequency of arrhythmias during serial exercise testing and clinical follow-up after Melody valve implant. Heart Rhythm. 2016 Nov;13(11):2135-2141. doi: 10.1016/j.hrthm.2016.07.023. Epub 2016 Jul 21. PMID 27453127
- [Derived] Cheatham JP, Hellenbrand WE, Zahn EM, Jones TK, Berman DP, Vincent JA, McElhinney DB. Clinical and hemodynamic outcomes up to 7 years after transcatheter pulmonary valve replacement in the US melody valve investigational device exemption trial. Circulation. 2015 Jun 2;131(22):1960-70. doi: 10.1161/CIRCULATIONAHA.114.013588. Epub 2015 May 5. PMID 25944758
- [Derived] McElhinney DB, Benson LN, Eicken A, Kreutzer J, Padera RF, Zahn EM. Infective endocarditis after transcatheter pulmonary valve replacement using the Melody valve: combined results of 3 prospective North American and European studies. Circ Cardiovasc Interv. 2013 Jun;6(3):292-300. doi: 10.1161/CIRCINTERVENTIONS.112.000087. Epub 2013 Jun 4. PMID 23735475
- [Derived] McElhinney DB, Cheatham JP, Jones TK, Lock JE, Vincent JA, Zahn EM, Hellenbrand WE. Stent fracture, valve dysfunction, and right ventricular outflow tract reintervention after transcatheter pulmonary valve implantation: patient-related and procedural risk factors in the US Melody Valve Trial. Circ Cardiovasc Interv. 2011 Dec 1;4(6):602-14. doi: 10.1161/CIRCINTERVENTIONS.111.965616. Epub 2011 Nov 9. PMID 22075927
- [Derived] McElhinney DB, Hellenbrand WE, Zahn EM, Jones TK, Cheatham JP, Lock JE, Vincent JA. Short- and medium-term outcomes after transcatheter pulmonary valve placement in the expanded multicenter US melody valve trial. Circulation. 2010 Aug 3;122(5):507-16. doi: 10.1161/CIRCULATIONAHA.109.921692. Epub 2010 Jul 19. PMID 20644013

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled: All subjects enrolled (n=171)
Period: Overall Study
Arm/Group | Enrolled
Started | 171
Completed | 150
Not Completed | 21
Not completed — Not Catheterized | 4
Not completed — Further testing contraindicated implant | 17

BASELINE CHARACTERISTICS:
Population: All stubjects enrolled
Groups:
- Enrolled Cohort: All subjects enrolled
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 107
Region of Enrollment [Number; unit: participants]
  United States | 171

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Freedom From TPV Dysfunction
Description: To assess whether long-term functionality of implantation of the Medtronic Melody TPV at 5 years is no worse than the historical control established through literature review. This study is designed to test the null hypothesis that the true freedom from TPV dysfunction at 5 years after Melody implantation (PMelody) is less than or equal to 36% (PControl). To reject the null hypothesis means that freedom from TPV dysfunction at 5 years after Melody implantation (PMelody) is greater than 36% (PControl). The null (H0) and alternative (HA) hypotheses are written as follows:H0: PMelody ≤ PControl and HA: PMelody > PControl. TPV dysfunction is a composite outcome defined as the following:
  * Hemodynamic dysfunction of the TPV
    * Moderate or greater pulmonary regurgitation, and/or
    * Mean Right Ventricular Outflow Tract (RVOT) gradient greater than 40 mmHg
  * RVOT reoperation for conduit dysfunction or device-related reasons
  * Catheter re-intervention on the TPV
Time Frame: 5 years
Population: The Implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Implanted >24 Hour Cohort: The Implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours.
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 72.9 [64.4 to 79.6]
Statistical Analysis 1: Comparison: Implanted >24 Hour Cohort; Test type: Superiority; p < 0.0001, Z test; Kaplan-Meier Rate = 74.2, 95% CI 1-sided [lower limit 67.1]

2. Secondary Outcome: Freedom From TPV Dysfunction at 10 Years
Description: The outcome measure for this objective is TPV dysfunction, which is a composite outcome defined as RVOT reoperation for conduit dysfunction or device-related reasons, catheter re-intervention on the TPV, or hemodynamic dysfunction of the TPV (moderate or greater pulmonary regurgitation, and/or a mean RVOT gradient greater than 40 mmHg).
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
Percentage of subjects | 52.9 [39.7 to 64.5]

3. Secondary Outcome: Procedural Success
Description: Procedural success is a composite outcome defined as:
  * Melody TPV fixated within the desired location
  * Right Ventricle (RV) - Pulmonary Artery (PA) peak-to-peak gradient (measured in the catheterization lab) less than 35 mmHg post-implant
  * Less than mild pulmonary regurgitation by angiography post-implant
  * Free of explant at 24 hours post-implant
Time Frame: Within 24 Hours post implant
Population: The attempted implant cohort consists of all subjects who underwent catheterization and a Melody TPV implantation was attempted (Melody TPV valve opened).
Measure: Number; unit: percentage of subjects
Groups:
- Attempted Implant Cohort: The attempted implant cohort consists of all subjects who underwent catheterization and a Melody TPV implantation was attempted (Melody TPV valve opened).
Arm/Group | Attempted Implant Cohort
Number analyzed (Participants) | 150
percentage of subjects | 94.7

4. Secondary Outcome: Serious Procedural Adverse Event (AE)
Description: A procedure-related event is defined as an event that is associated with the implant procedure by the chronology or physiology and was caused by the implant procedure (e.g. rupture of the conduit or damage to an intra-cardiac or intravascular structure by the delivery system).
Time Frame: 5 years
Population: The catheterized cohort consists of all subjects who underwent catheterization for possible implantation of the Melody TPV.
Measure: Number; unit: Percent of subjects
Groups:
- Catheterized Cohort: The catheterized cohort consists of all subjects who underwent catheterization for possible implantation of the Melody TPV.
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 167
Percent of subjects | 12.6

5. Secondary Outcome: Serious Procedural Adverse Event (AE)
Description: as for outcome 4
Time Frame: 10 years
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 167
percentage of subjects | 13.2

6. Secondary Outcome: Serious Device-related Adverse Event
Description: A device-related event is defined as an event that is associated with the TPV by the chronology or physiology and was caused by the the TPV (e.g. embolization of the TPV and any adverse events which follow).
Time Frame: 5 years
Population: The implanted cohort consists of all subjects who underwent catheterization and a Melody TPV was implanted.
Measure: Number; unit: Percentage of subjects
Groups:
- Implanted Cohort: The implanted cohort consists of all subjects who underwent catheterization and a Melody TPV was implanted.
Arm/Group | Implanted Cohort
Number analyzed (Participants) | 150
Percentage of subjects | 28

7. Secondary Outcome: Serious Device-related Adverse Event
Description: as for outcome 6
Time Frame: 10 years
Population: The implanted cohort consists of all subjects who underwent catheterization and a Melody TPV was implanted.
Measure: Number; unit: percentage of subjects
Arm/Group | Implanted Cohort
Number analyzed (Participants) | 150
percentage of subjects | 41.3

8. Secondary Outcome: Kaplan-Meier Freedom From Major Stent Fracture at 5 Years
Description: Major stent fracture is defined as a stent fracture requiring intervention to prevent permanent impairment of a body function or permanent damage to a body structure.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 84.3 [72.8 to 91.2]

9. Secondary Outcome: Kaplan-Meier Freedom From Major Stent Fracture at 10 Years
Description: as for outcome 8
Time Frame: 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 83.7 [69.8 to 91.6]

10. Secondary Outcome: Kaplan-Meier Freedom From Catheter Re-intervention on TPV
Description: Catheter Re-intervention is defined as: any catheter-based intervention involving the TPV, including balloon dilatation, stenting, or placement of a second TPV
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 81 [72.9 to 86.9]

11. Secondary Outcome: Kaplan-Meier Freedom From Catheter Re-intervention on TPV
Description: as for outcome 10
Time Frame: 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 73.1 [58.4 to 83.3]

12. Secondary Outcome: Kaplan-Meier Freedom From Surgical Replacement of the RVOT Conduit
Description: Surgical Replacement of the RVOT Conduit is defined as any surgical procedure to repair, alter, or explant the TPV
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 92.2 [86.2 to 95.7]

13. Secondary Outcome: Kaplan-Meier Freedom From Surgical Replacement of the RVOT Conduit
Description: Surgical Replacement of the RVOT Conduit is defined as any surgical procedure to repair, alter, or explant the TPV
Time Frame: 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 149
percentage of subjects | 78.9 [66.5 to 87.1]

14. Secondary Outcome: Kaplan-Meier Freedom From Death (All-cause, Procedural and Device-related)
Description: Deaths is defined as all-cause, procedural and device-related events at 5 years
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 167
percentage of subjects | 96.5 [91.4 to 98.6]

15. Secondary Outcome: Kaplan-Meier Freedom From Death (All-cause, Procedural and Device-related)
Description: Deaths is defined as all-cause, procedural and device-related events at 10 years
Time Frame: 10 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 167
percentage of subjects | 90.2 [78.5 to 95.7]

16. Secondary Outcome: Functional Assessment (NYHA Classification)
Description: Improvement in Functional Assessment (NYHA Classification) at 6 months post implant.
Time Frame: 6 Months
Population: The Implanted >24 hours cohort consists of all subjects who had a Melody TPV implanted which remained implanted for greater than 24 hours and had paired data from pre-implant to 6 months post-implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted >24 Hour Cohort
Number analyzed (Participants) | 143
Participants
  Improved | 102
  No Change | 39
  Worsened | 1
  Died | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent through end of participation in the study.
Description: Any undesirable clinical occurrence or untoward deviation in health from the patient's baseline condition at the time of consent. Clinically significant worsening of a baseline condition requiring a new intervention, Deterioration of primary disease, Intercurrent illness, AEs related or possibly related to the implant that are greater in intensity and require different clinical intervention than normally required, and Abnormal findings on diagnostic tests not present at the onset of the study.
Arm/Group | Catheterized Cohort
All-Cause Mortality (participants affected / at risk) | 8/167
Serious Adverse Events (participants affected / at risk) | 106/167
Other Adverse Events (participants affected / at risk) | 112/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=167)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Aortic Regurgitation (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrial Flutter (Cardiac disorders) | 9 (13)
Cardiac Arrest (Cardiac disorders) | 4 (4)
Cardiac Disorder (Cardiac disorders) | 11 (13)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 4 (7)
Intracardiac Mass (Cardiac disorders) | 1 (2)
Premature Ventricular Ectopic Beats (Cardiac disorders) | 2 (2)
Pulmonary Valve Disease (Cardiac disorders) | 2 (2)
Pulmonary Valve Regurgitation (Cardiac disorders) | 3 (3)
Pulmonary Valve Stenosis (Cardiac disorders) | 33 (56)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid Regurgitation (Cardiac disorders) | 5 (8)
Ventricular Fibrillation (Cardiac disorders) | 2 (3)
Ventricular Tachycardia (Cardiac disorders) | 10 (12)
Gastrointestinal Disorder (Gastrointestinal disorders) | 4 (5)
Other Events (General disorders) | 15 (23) — For the 23 "other serious" events reported by the sites as "other" event, the only event reported >once was depression (3 subjects). All the rest were unique events.
Chest Pain (General disorders) | 3 (4)
Device Complication (General disorders) | 10 (10)
Device Rupture (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Multi Organ Failure (General disorders) | 2 (2)
Prosthetic Cardiac Valve Malfunction (General disorders) | 1 (1)
Prosthetic Tissue Defect (General disorders) | 1 (1)
Stent Strut Fracture (General disorders) | 23 (28)
Endocarditis (Infections and infestations) | 11 (18)
Infection (Infections and infestations) | 8 (11)
Pneumonia (Infections and infestations) | 2 (2)
Prosthetic Valve Endocarditis (Infections and infestations) | 18 (33)
Sepsis (Infections and infestations) | 9 (9)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Procedural Complication (Injury, poisoning and procedural complications) | 2 (2)
Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (2)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Prosthetic Cardiac Valve Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Central Nervous System Disorder (Nervous system disorders) | 4 (4)
Cva (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (5)
Acute Renal Failure (Renal and urinary disorders) | 3 (3)
Renal Disorder (Renal and urinary disorders) | 1 (2)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Thromboembolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Vascular Dissection (Vascular disorders) | 1 (1)
Venous Thrombosis (Vascular disorders) | 1 (2)
Vessel Perforation (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=167)
Hemolysis (Blood and lymphatic system disorders) | 9 (15)
Arrhythmia (Cardiac disorders) | 10 (12)
Cardiac Disorder (Cardiac disorders) | 16 (18)
Palpitations (Cardiac disorders) | 16 (23)
Tricuspid Regurgitation (Cardiac disorders) | 12 (14)
Gastrointestinal Disorder (Gastrointestinal disorders) | 9 (9)
Other Events (General disorders) | 35 (69) — For the 69 "other" events reported by the sites as "other" event, the only events reported >twice were fatigue (5), depression (4), anxiety (4) and abdominal pain (3)
Chest Pain (General disorders) | 17 (25)
Stent Strut Fracture (General disorders) | 51 (73)
Infection (Infections and infestations) | 9 (15)
Central Nervous System Disorder (Nervous system disorders) | 9 (10)
Headache (Nervous system disorders) | 11 (16)
Renal Disorder (Renal and urinary disorders) | 14 (29)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 16 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days